CLINICAL TRIAL: NCT06790030
Title: Does Self-Efficacy at the Start of Treatment Predict Treatment Outcome in Patients With EDs?
Brief Title: Does Self-Efficacy at the Start of Treatment Influence Treatment Outcome in Patients With EDs?
Status: Recruiting | Type: Observational
Sponsor: Altrecht (Other)
Responsible Party: Principal Investigator, Alberte Jansingh, Clinical psychologist; Lead Expert Eatingdisorders Altrecht, Altrecht
Other Study IDs: CWO-nr2227
Record Dates: First submitted 2024-11-27; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Eating Disorders
Keywords: treatment; self-efficacy
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: CBT-T — cognitive behavioral therapy-ten :

SUMMARY:
The goal of this clinical trial is to contribute to the improvement of treatment for eating disorders, by identifying factors that might positively affect treatment outcome.

The main questions it aims to answer are:

1. Do higher levels of self-efficacy positively predict a more positive treatment outcome?
2. Does self-efficacy in itself improve during treatment?
3. Do autonomous motivation, self-esteem and self-efficacy correlate?

These factors will be measured in patients being treated for their eating disorders with Cognitive Behavior Therapy - Ten (CBT-T).

Researchers will administer questionnaires at start, session four and end of treatment.

Participants will:

1. Receive their treatment as usual.
2. fill in questionnaires at the start of treatment, session 4 and end of treatment.

DETAILED DESCRIPTION:
Eating disorders (EDs) are severe psychiatric disorders, characterized by a persistent disturbance of eating which impairs health or psychosocial functioning and causes loss of quality of life. There are several evidence-based forms of treatment, but outcomes are mediocre at best. Previous research found better treatment outcomes with several baseline predictors, such as greater motivation to recover. Research on motivation to change has indicated that autonomous motivated (AM) individuals show better response to treatments for EDs. However, being highly motivated for change, but not experiencing the capacity to really eat more and to deal with the emotions evoked by the process of recovery, might lead to difficulty to change key-behaviors, thus leading to less positive treatment outcome. Several researchers emphasized the importance of self-efficacy as a predictor in eating attitudes and behaviors. This study focuses on whether self-efficacy at the start of treatment is predictive of treatment outcome, measured by the ED-15 questionnaire in patients with an ED. Data will be obtained during CBT-T; a brief (10 sessions) version of cognitive behavioral therapy for eating disorders like BN, BED and OSFED. In CBT-T patients are encouraged, from the start of treatment, to challenge their fears, experience the effect of exposure and motivating them to carry through. This aspect might enlarge patients' experience of self-efficacy. Patients with low level of self-efficacy at start, but higher level of self-efficacy after four sessions, might benefit better from treatment, then patients with lower levels of self-efficacy throughout the treatment. To study this potential effect of treatment on self-efficacy, self-efficacy will be measured at start of treatment, at session four and at the end of treatment.

Self-efficacy, self-esteem and autonomous motivation are concepts that are closely linked to each other. To test if they are positively correlated at start of treatment, measurements covering these concepts will be included at T0.

HYPOTHESES

Primary hypotheses:

Higher levels of self-efficacy will positively predict a more positive treatment outcome as determined by lower eating pathology levels with the ED-15.

Secondary hypotheses:

1. Self-efficacy in itself will improve during treatment.
2. Autonomous motivation, self-esteem and self-efficacy will be positively correlated.

ELIGIBILITY:
Patients are eligible for participation when they meet the following inclusion criteria:

* Participants must be 18 years or older
* Having an eating disorder diagnosed according to the Diagnostic Statistical Manual (DSM-5)
* Starting CBT-T treatment

Exclusion criteria

* Intellectual disability according to the Diagnostic Statistical Manual (DSM-5) or an IQ below 80
* Inability to speak or read Dutch
* Patients treated under a legal act

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (adult) Patients treated for eatingdisorders with CBT-T at Altrecht Eating Disorders Rintveld or at Co-eur.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
treatment outcome | CBT-T is a weekly, ten-session treatment. The ED-15 will be adminstered at the start of the first treatment session, at session 4 and at the end of treatment (session 10).: * week 1 * week 4 * week 10
  Eating Disorder-15 (ED-15) is a self-report questionnaire used to measure session-by-session change in eating pathology as part of the CBT-T protocol. All items are positively scored from 0-6, with higher scores reflecting higher levels of eating disorder pathology.

SECONDARY OUTCOMES:
General Self-efficacy | CBT-T is a weekly, ten-session treatment. The GSES will be adminstered at at the start of the first treatment session , at session 4 and at the end of treatment (session 10): * week 1 * week 4 * week 10
  Dutch General Self-Efficacy Scale (GSES) 10 item self-report to measure self-efficacy. four-point Likert scale, ranging from not at all true (1) to exactly true (4). The total score is calculated by finding the sum of all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Coping Self-efficacy | CBT-T is a weekly, ten-session treatment. The CSES will be adminstered at the start of the first treatment session , at session 4 and at the end of treatment (session 10): * week 1 * week 4 * week 10
  Coping Self-Efficacy Scale (CSES) The CSES is a 26-item measure of one's confidence in performing coping behavior when facing life challenges. 11-point Likert scale : 0 - "cannot do at all", 5 - "moderately certain can do", and 10 - "certain can do. Item scores are summated to create an overall CSES score (maximum 260). The higher the score, the higher the level of coping self-efficacy

OTHER OUTCOMES:
Autonomous motivation | CBT-T is a weekly, ten-session treatment. The ACMTQ will be adminstered at the start of the first treatment session: *week 1
  Autonomous and Controlled Motivation for Treatment Questionnaire (ACMTQ) - Dutch Translation, adjusted to ED population by replacing the word depression to eating disorders.
  The seven-point Likert scale ranges from 1 (strongly disagree) to 7 (strongly agree). Two mean scores are derived, one per subscale. Higher scores indicate stronger endorsement of the motivation type.
Self-esteem | CBT-T is a weekly, ten-session treatment. The RSES will be adminstered at the start of the first treatment session: *week 1
  Rosenberg Self-Esteem Scale (RSES), 10-item scale, four-point Likert scale format, ranging from strongly agree to strongly disagree. Higher scores indicate higher self-esteem.
Motivation | CBT-T is a weekly, ten-session treatment. The Motivational Ruler will be adminstered at the start of the first treatment session: * week 1.
  Motivational Ruler Identifies the ability to change and importance to change; range 0-10). Higher scores reflect a higher motivation to change.

CONTACTS AND LOCATIONS:
Locations (1):
- Altrecht Eatings Disorders Rintveld, Zeist, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
data will be profided in case of a specific request. Data will be stored anonymously in a database on a special drive for scientific research at Altrecht. Researchers will act according to the Declaration of Helsinki, version 59th WMA General Assembly, October 2008. All study data will be stored in a coded way and the key-to-the-name information will be stored in a separate file which will only be accessible to researchers directly involved in the study. The data will be handled confidently and anonymously and will be stored for at least 15 years, in line with the article 454 section 3 from "Wet op de Geneeskundige Behandelingsovereenkomst - WGBO". Only the researchers who are directly involved in this project will have access to the data. The data will be described at group level. All data will be handled and described within the Altrecht workspace.
Supporting Information: Study Protocol, ICF
Time Frame: for the next 15 years
Access Criteria: information can be obtained by contacten the researchers.

REFERENCES:
- [Background] Denison-Day J, Appleton KM, Newell C, Muir S. Improving motivation to change amongst individuals with eating disorders: A systematic review. Int J Eat Disord. 2018 Sep;51(9):1033-1050. doi: 10.1002/eat.22945. Epub 2018 Sep 6. PMID 30189116
- [Background] Waller G, Tatham M, Turner H, Mountford VA, Bennetts A, Bramwell K, Dodd J, Ingram L. A 10-session cognitive-behavioral therapy (CBT-T) for eating disorders: Outcomes from a case series of nonunderweight adult patients. Int J Eat Disord. 2018 Mar;51(3):262-269. doi: 10.1002/eat.22837. Epub 2018 Feb 8. PMID 29417603
- [Background] Tatham M, Turner H, Mountford VA, Tritt A, Dyas R, Waller G. Development, psychometric properties and preliminary clinical validation of a brief, session-by-session measure of eating disorder cognitions and behaviors: The ED-15. Int J Eat Disord. 2015 Nov;48(7):1005-15. doi: 10.1002/eat.22430. Epub 2015 May 26. PMID 26011054
- [Background] Steiger H, Sansfacon J, Thaler L, Leonard N, Cottier D, Kahan E, Fletcher E, Rossi E, Israel M, Gauvin L. Autonomy support and autonomous motivation in the outpatient treatment of adults with an eating disorder. Int J Eat Disord. 2017 Sep;50(9):1058-1066. doi: 10.1002/eat.22734. Epub 2017 Jun 14. PMID 28842966
- [Background] Steele AL, Bergin J, Wade TD. Self-efficacy as a robust predictor of outcome in guided self-help treatment for broadly defined bulimia nervosa. Int J Eat Disord. 2011 Jul;44(5):389-96. doi: 10.1002/eat.20830. Epub 2010 Aug 18. PMID 20721895
- [Background] Sansfacon J, Fletcher E, Zuroff DC, Schmitz N, Miller A, Israel M, Steiger H. Psychometric properties of the "Autonomous and Controlled Motivation for Treatment Questionnaire" in women with eating disorders. Eur Eat Disord Rev. 2019 May;27(3):306-314. doi: 10.1002/erv.2656. Epub 2018 Nov 12. PMID 30417472
- [Background] Mansour S, Bruce KR, Steiger H, Zuroff DC, Horowitz S, Anestin AS, Sycz L. Autonomous motivation: a predictor of treatment outcome in bulimia-spectrum eating disorders. Eur Eat Disord Rev. 2012 May;20(3):e116-22. doi: 10.1002/erv.2154. Epub 2012 Feb 7. PMID 22311824
- [Background] Linardon J, de la Piedad Garcia X, Brennan L. Predictors, Moderators, and Mediators of Treatment Outcome Following Manualised Cognitive-Behavioural Therapy for Eating Disorders: A Systematic Review. Eur Eat Disord Rev. 2017 Jan;25(1):3-12. doi: 10.1002/erv.2492. Epub 2016 Nov 16. PMID 27862611
- [Background] Hasking P, Boyes M, Greves S. Self-efficacy and emotionally dysregulated behaviour: An exploratory test of the role of emotion regulatory and behaviour-specific beliefs. Psychiatry Res. 2018 Dec;270:335-340. doi: 10.1016/j.psychres.2018.09.045. Epub 2018 Sep 20. PMID 30292086
- [Background] Hamadi L, Holliday J. Moderators and mediators of outcome in treatments for anorexia nervosa and bulimia nervosa in adolescents: A systematic review of randomized controlled trials. Int J Eat Disord. 2020 Jan;53(1):3-19. doi: 10.1002/eat.23159. Epub 2019 Sep 11. PMID 31506978
- [Background] Eisenberg MH, Lipsky LM, Dempster KW, Liu A, Nansel TR. I Should but I Can't: Controlled Motivation and Self-Efficacy Are Related to Disordered Eating Behaviors in Adolescents With Type 1 Diabetes. J Adolesc Health. 2016 Nov;59(5):537-542. doi: 10.1016/j.jadohealth.2016.06.008. Epub 2016 Aug 23. PMID 27567063
- [Background] Clarke J, Proudfoot J, Birch MR, Whitton AE, Parker G, Manicavasagar V, Harrison V, Christensen H, Hadzi-Pavlovic D. Effects of mental health self-efficacy on outcomes of a mobile phone and web intervention for mild-to-moderate depression, anxiety and stress: secondary analysis of a randomised controlled trial. BMC Psychiatry. 2014 Sep 26;14:272. doi: 10.1186/s12888-014-0272-1. PMID 25252853
- [Background] Chesney MA, Neilands TB, Chambers DB, Taylor JM, Folkman S. A validity and reliability study of the coping self-efficacy scale. Br J Health Psychol. 2006 Sep;11(Pt 3):421-37. doi: 10.1348/135910705X53155. PMID 16870053
- [Background] Chang PGRY, Delgadillo J, Waller G. Early response to psychological treatment for eating disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2021 Jun;86:102032. doi: 10.1016/j.cpr.2021.102032. Epub 2021 Apr 18. PMID 33915335
- [Background] Bruijniks SJ, Bosmans J, Peeters FP, Hollon SD, van Oppen P, van den Boogaard M, Dingemanse P, Cuijpers P, Arntz A, Franx G, Huibers MJ. Frequency and change mechanisms of psychotherapy among depressed patients: study protocol for a multicenter randomized trial comparing twice-weekly versus once-weekly sessions of CBT and IPT. BMC Psychiatry. 2015 Jun 30;15:137. doi: 10.1186/s12888-015-0532-8. PMID 26122891
- [Background] Bosscher RJ, Smit JH. Confirmatory factor analysis of the General Self-Efficacy Scale. Behav Res Ther. 1998 Mar;36(3):339-43. doi: 10.1016/s0005-7967(98)00025-4. PMID 9642852
- [Background] Bardone-Cone AM, Thompson KA, Miller AJ. The self and eating disorders. J Pers. 2020 Feb;88(1):59-75. doi: 10.1111/jopy.12448. Epub 2018 Dec 30. PMID 30506587